CLINICAL TRIAL: NCT01418716
Title: A Program to TRANSform InTerprofessional Clinical Practices to Improve Cardiovascular Prevention in Primary Care
Brief Title: TRANSforming InTerprofessional Cardiovascular Prevention in Primary Care
Acronym: TRANSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonds de la Recherche en Santé du Québec (Other Government)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Lyne Lalonde, Professor (professeur agrégé), Fonds de la Recherche en Santé du Québec
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FRSQ-22424
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Cholesterol, LDL; Comorbitdity
Keywords: Disease Management; Quality Improvement; Cooperative Behavior (collaboration)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Cooperative Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facilitation (Experimental): Facilitation is a change management process. In the TRANSIT study, the change consist in implementing the TRANSIT program in primary care clinics. In the facilitation group, external facilitators accompany, support, and empower clinical teams so they quickly develop a sense of ownership regarding new clinical practices and sustainably implement them with lower costs. External facilitators offer counseling, coaching, and various tools to an internal facilitation team composed of clinicians of the clinical team to support their efforts in implementing change in their practices. Facilitation activities are structured in a cycle of 4 steps, the Plan-Do-Study-Act cycle (PDSA cycle).
  Interventions: Other: Facilitation
- Passive diffusion (Active Comparator): Clinical teams in primary care clinics implement the TRANSIT program without the help of facilitators.
  Interventions: Other: Passive diffusion

INTERVENTIONS:
Other: Facilitation — Facilitation is a change management process. In the TRANSIT study, the change consist in implementing the TRANSIT program in primary care clinics. In the facilitation group, external facilitators accompany, support, and empower clinical teams so they quickly develop a sense of ownership regarding new clinical practices and sustainably implement them with lower costs. External facilitators offer counseling, coaching, and various tools to an internal facilitation team composed of clinicians of the clinical team to support their efforts in implementing change in their practices. Facilitation activities are structured in a cycle of 4 steps, the Plan-Do-Study-Act cycle (PDSA cycle).
  Other Names: Plan-Do-Study-Act cycles (PDSA cycles)
  Arms: Facilitation
Other: Passive diffusion — Clinical teams in primary care clinics implement the TRANSIT program without the help of facilitators.
  Arms: Passive diffusion

SUMMARY:
The TRANSIT program is a program to TRANSform InTerprofessional clinical practices to improve cardiovascular prevention in primary care. It addresses priorities in primary care relevant to the Chronic Care Model (Wagner 2001): self-management support, delivery-system design, and management of clinical information.

The program includes :

* a case manager to coordinate and provide care and follow up;
* clinical protocols and tools to support interprofessional and systematic follow up;
* training for clinicians;
* patient's personalized cardiovascular health booklet;
* tools to promote group sessions for patient education on cholesterol, hypertension, and diabetes.

The general OBJECTIVE of this trial is to evaluate and compare two STRATEGIES for implementing the TRANSIT program in Family Medicine Groups (FMGs):

1. facilitation, and
2. passive diffusion.

Passive diffusion is the usual strategy where clinicians implement an intervention program by themselves. Facilitation is a strategy whereby a facilitator provides support to a team of clinicians to help them introduce the changes required to implement the program into practice.

The hypothesis is that facilitation will be more efficacious to implement the program than passive diffusion:

* it will enhance the provision of cardiovascular preventive care;
* it will enhance interprofessional collaboration;
* it will enable more efficaciously the implementation of new clinical processes;
* it will improve patient clinical outcomes;
* it will cost more in the short term, but will have positive economic impact in the long term;
* there will be less "undesired effects" of all types related to implementation.

To test the hypothesis, we assess the efficacy of the implementation strategies to enhance interprofessional collaboration and better support patients in the management of their conditions. Impact on provision of care, interprofessional collaboration, clinical processes, and patient clinical outcomes (values, therapeutic targets, and lifestyle habits) will be evaluated. Moreover, the implementation cost related to each strategy will be estimated.

We complement the trial with qualitative methods to document the perceptions of clinicians, facilitators, patients and members of the family regarding the TRANSIT program, the implementation strategies and the observed changes in the clinical practices and outcomes.

DETAILED DESCRIPTION:
STUDY DESIGN:

Pragmatic cluster randomized clinical trial

SETTING:

Nine Family Medicine Groups (FMGs) take part in the study. FMGs are primary care clinics delivering family medicine services. They include physicians and nurses, and collaborate with other health professionals.

Eligible FMGs meet the following criteria:

1. 2 physicians, 1 nurse, 1 community pharmacist, 1 member of the medical administrative support, and 1 other health professional (nutritionist, kinesiologist, or psychologist) accept to participate by collaborating to the facilitation activities, if the FMG is assigned to the facilitation group;
2. 1 physician, 1 nurse, 1 community pharmacist and 1 other health professional (nutritionist, psychologist, kinesiologist) accept to play a role in the internal facilitation team, if the FMG is assigned to the facilitation group;
3. a room is available for the case manager nurse for the equivalent of one day/week over 15 months;
4. 100 eligible patients accept to participate in the study, with a minimum of 15 patients per physician participant.

All FMGs in the TRANSIT study are given access to the TRANSIT program, to the supportive clinical tools cliniques, and to a case manager nurse. Training will be offered on the use of the electronic directory of health resources and on motivational interview.

RANDOMIZATION:

Prior to randomization, each clinician is assigned to one FMG only. Each FMG will be paired with 2 others of the same level of CVD preventive care (score <6 or ≥6), as estimated with the questionnaire "Assessment of Chronic Illness Care" (ACIC). Usually, medical clinics report a score of 5 or less at baseline.

Participating FMGs (n=9) will be randomly assigned to facilitation (n=6) and to passive diffusion (n=3). FMGs will be randomized simultaniously in blocs of 3. For each bloc, 2:1 ratio (facilitation:passive diffusion) will be respected. Randomization will be stratified in fonction of the ACIC score (score <6 or score ≥6). Because of the small number of participating FMGs, grouping GMFs in blocs of 3 according to the ACIC score will ensure complete blocs are found in each randomization stratum.

ANALYSIS:

For all variables, multivariable analysis models taking account the intracluster correlation (linear/SAS PROC MIXED) for continuous and categorical variables (logistic/PROC GENMOD) will be developed. Significative variables (p<0.2) in bivariable model including the study group will be included in the multivariable model. We will then apply a backward selection procedure and include in the final model those variables that were statistically significant at p < 0.1.

ELIGIBILITY:
Inclusion Criteria:

* patient is registered in a Family Medicine Group;
* 10-year Framingham risk score (FRS) moderate (11-19%) to high (≥ 20%);
* at least one of the following condition uncontrolled:

  * Diabetes: HbA1C > 7% OR fasting blood glucose > 7 mmol/L OR 2-hour postprandial blood glucose > 10 mmol/L (OR > 8 mmol/L if HbA1C target is not acheived)(Canadian Diabetes Association Clinical Practice Guidelines Expert Committee, Canadian Journal of Diabetes, 2008)
  * Dyslipidemia: C-LDL ≥ 2 mmol/L in moderate to high risk patients OR less than 50% reduction of C-LDL compared to initial value OR Apo-B ≥ 0,8 g/L (Genest, McPherson et al. 2009)
  * Hypertension: blood pressure ≥ 140/90 ou ≥ 130/80 in diabetic patients or with chronic kidney disease (TFG < 60mL/min/1,73m2; (Cloutier & Poirier 2011)
* Patient with at least two chronic disease or chronic health problem other than type II diabetes, dyslipidemia, hypertension, or cardiovascular disease (e.g. : angina, previous history of myocard infarct, stroke, and intermittent claudication).

Exclusion Criteria:

* Patient followed for a cardiovascular disease in a specialized clinic in secondary care (ex.: cardiology, endocrinology etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Quality of the cardiovascular preventive care | Baseline and 12 months after randomization
  Mean change in the composite score of the quality of the cardiovascular preventive care

SECONDARY OUTCOMES:
Organisational outcomes | Baseline and 12 months after randomization
  Impact of implementation strategy on:
  1. clinicians' and patients' perception of health service delivery (questionnaires: ACIC and PACIC);
  2. team work (questionnaire: TCI - short version);
  3. clinicians' perception of achievement of change (questionnaires: Herscovitch and Meyer's Affective Engagement, Bandura's Self Efficacy, and clinician's perception of achievement of the TRANSIT program [after 12 months only]);
  4. direct costs (clinician time and compensations for participation in facilitation activities, salary and training of the external facilitator).
Blood pressure | Baseline and 12 months after randomization
  Mean change in the systolic/diastolic blood pressure
c-LDL | Baseline and 12 months after randomization
  Mean change in change in the c-LDL
Glycosylated hemoglobine (HgA1c) | Baseline and 12 months after randomization
  Mean change in the HgA1c
Achieved therapeutic targets | Baseline and 12 months after randomization
  Mean change in percentage of achieved therapeutic targets
Lifestyle habits | Baseline and 12 months after randomization
  Mean change in lifestyle habits as measured using self-administered questionnaires to patients : Hopkin's food frequency questionnaire, International Physical Activity Questionnaire (IPAQ), smoking status
Use of public programs | Baseline and 12 months after randomization
  Mean change in percentage of patients using the education programs and in mean frequency of use. Programs are education to patients on diabetes, cholesterol, hypertension, and healthy weight control

CONTACTS AND LOCATIONS:
Overall Officials: Lyne Lalonde, Ph.D., Principal Investigator — Centre de santé et de services sociaux de Laval ; University of Montreal; Johanne Goudreau, Ph.D., Principal Investigator — Université de Montréal; Céline Bareil, Ph.D., Principal Investigator — HEC Montréal; Éveline Hudon, M.D., Principal Investigator — Université de Montréal; Fabie Duhamel, Ph.D., Principal Investigator — Université de Montréal; Marie-Thérèse Lussier, M.D., Principal Investigator — Université de Montréal
Locations (1):
- Centre de santé et de services sociaux de Laval, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Background] Dogherty EJ, Harrison MB, Graham ID. Facilitation as a role and process in achieving evidence-based practice in nursing: a focused review of concept and meaning. Worldviews Evid Based Nurs. 2010 Jun 1;7(2):76-89. doi: 10.1111/j.1741-6787.2010.00186.x. Epub 2010 Feb 19. PMID 20180826
- [Background] Nagykaldi Z, Mold JW, Robinson A, Niebauer L, Ford A. Practice facilitators and practice-based research networks. J Am Board Fam Med. 2006 Sep-Oct;19(5):506-10. doi: 10.3122/jabfm.19.5.506. PMID 16951300
- [Background] Genest J, McPherson R, Frohlich J, Anderson T, Campbell N, Carpentier A, Couture P, Dufour R, Fodor G, Francis GA, Grover S, Gupta M, Hegele RA, Lau DC, Leiter L, Lewis GF, Lonn E, Mancini GB, Ng D, Pearson GJ, Sniderman A, Stone JA, Ur E. 2009 Canadian Cardiovascular Society/Canadian guidelines for the diagnosis and treatment of dyslipidemia and prevention of cardiovascular disease in the adult - 2009 recommendations. Can J Cardiol. 2009 Oct;25(10):567-79. doi: 10.1016/s0828-282x(09)70715-9. PMID 19812802
- [Background] Hackam DG, Khan NA, Hemmelgarn BR, Rabkin SW, Touyz RM, Campbell NR, Padwal R, Campbell TS, Lindsay MP, Hill MD, Quinn RR, Mahon JL, Herman RJ, Schiffrin EL, Ruzicka M, Larochelle P, Feldman RD, Lebel M, Poirier L, Arnold JM, Moe GW, Howlett JG, Trudeau L, Bacon SL, Petrella RJ, Milot A, Stone JA, Drouin D, Boulanger JM, Sharma M, Hamet P, Fodor G, Dresser GK, Carruthers SG, Pylypchuk G, Burgess ED, Burns KD, Vallee M, Prasad GV, Gilbert RE, Leiter LA, Jones C, Ogilvie RI, Woo V, McFarlane PA, Hegele RA, Tobe SW; Canadian Hypertension Education Program. The 2010 Canadian Hypertension Education Program recommendations for the management of hypertension: part 2 - therapy. Can J Cardiol. 2010 May;26(5):249-58. doi: 10.1016/s0828-282x(10)70379-2. PMID 20485689
- [Background] Fortin M, Soubhi H, Hudon C, Bayliss EA, van den Akker M. Multimorbidity's many challenges. BMJ. 2007 May 19;334(7602):1016-7. doi: 10.1136/bmj.39201.463819.2C. PMID 17510108
- [Background] Lalonde L, Goudreau J, Hudon E, Lussier MT, Duhamel F, Belanger D, Levesque L, Martin E; Group for TRANSIT to Best Practices in Cardiovascular Disease Prevention in Primary Care. Priorities for action to improve cardiovascular preventive care of patients with multimorbid conditions in primary care--a participatory action research project. Fam Pract. 2012 Dec;29(6):733-41. doi: 10.1093/fampra/cms021. Epub 2012 Feb 29. PMID 22379187
- [Background] Lalonde L, Goudreau J, Hudon E, Lussier MT, Bareil C, Duhamel F, Levesque L, Turcotte A, Lalonde G; Group for TRANSIT to Best Practices in Cardiovascular Disease Prevention in Primary Care. Development of an interprofessional program for cardiovascular prevention in primary care: A participatory research approach. SAGE Open Med. 2014 Feb 17;2:2050312114522788. doi: 10.1177/2050312114522788. eCollection 2014. PMID 26770705
- See also: Protocole de suivi interprofessionnel TRANSIT et outils cliniques associés (in French only) — http://www.recherchepl.ca/autres-productions-scientifiques.php